CLINICAL TRIAL: NCT02067429
Title: Limbal Relaxing Incisions Versus Toric Intraocular Lens for Keratometric Astigmatism <2.5 Diopters in Patients Undergoing Cataract Surgery and Intraocular Lens Implantation.
Brief Title: Limbal Relaxing Incision Versus Toric Intraocular Lens for Corneal Astigmatism During Cataract Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christin Henein (Other Government)
Collaborators: Rayner Intraocular Lenses Limited (Industry)
Responsible Party: Sponsor-Investigator, Christin Henein, Academic Foundation Doctor, Sussex Eye Hospital
Organization: Sussex Eye Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCT135670
Record Dates: First submitted 2014-02-17; First posted 2014-02-20 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Astigmatism; Cataract
MeSH Terms: conditions — Astigmatism; Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Toric Intraocular lens (Experimental): Toric intraocular lens implantation during standard cataract surgery
  Interventions: Device: Toric Intraocular Lens
- Limbal Relaxing Incisions (Experimental): Limbal relaxing incisions during standard cataract surgery
  Interventions: Procedure: Limbal Relaxing Incisions

INTERVENTIONS:
Procedure: Limbal Relaxing Incisions
  Arms: Limbal Relaxing Incisions
Device: Toric Intraocular Lens
  Arms: Toric Intraocular lens

SUMMARY:
This study will compare toric intra-ocular lens (IOL) with limbal relaxing incisions (LRI) in correcting astigmatism in patient undergoing standard cataract surgery.

Astigmatism is unequal curvature of the eye; the eye is oval rather than spherical. Uncorrected astigmatism of greater than approximately 0.75 diopters (D) can cause visual blurring, ghosting of images or halos. Over 20% of patients undergoing cataract surgery have astigmatism which is likely to have been corrected by spectacles.

Cataract surgery involves the replacement of the natural opacifying crystalline lens with a clear artificial plastic intra-ocular lens (IOL). The lens power can be selected to correct the patient's glasses prescription. The most widely used IOLs only correct glasses at one distance i.e. either near or distance. Residual astigmatism after cataract surgery will need glasses for correction which is undesirable for many patients.

Limbal relaxing incisions (LRI) are circumferential partial thickness cuts to the clear window of the eye (cornea) during surgery. These LRIs can correct corneal astigmatism and have no additional risk of complications.

Alternatively, toric IOLs are available which correct astigmatism inside the eye. They have been available for routine use in the last few years; technology has markedly improved and the lenses have become cheaper.

Studies have suggested toric IOLs provide better vision after cataract surgery than the regular IOLs. Toric IOL are widely used in the private practice and increasingly in the National Health Service (NHS). LRIs are cost effective for treating astigmatism however their predictability is believed to be lower than toric IOLs. As there are no randomised controlled trials comparing the outcomes between LRIs and toric IOLs. This research will address this gap in knowledge and accordingly from this research future practice will be able to provide treatment to patients with information about the best outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic cataract for which the patient desires surgery
2. Corneal astigmatism of greater than or equal to 0.75 D and lesser than or equal to 2.5D.
3. No significant ophthalmic co-morbidity which would affect the postoperative visual outcomes.

Exclusion Criteria:

1. <18 years of age
2. Significant ophthalmic comorbidity detrimental to final visual outcomes
3. Not competent to give consent
4. Concurrent use of ocular medications including lubricants
5. Unable to attend follow ups at 1, 3, 6 and 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Unaided distance LogMAR visual acuity (UDVA) | 1 months
Unaided distance LogMAR visual acuity (UDVA) | 3 months
Unaided distance LogMAR visual acuity (UDVA) | 6 months
Unaided distance LogMAR visual acuity (UDVA) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sussex Eye Hospital, Brighton, United Kingdom